CLINICAL TRIAL: NCT06819462
Title: Inhalaed Polymyxin E to Prevent Ventilator-associated Pneumonia: a Multicenter Clinical Study
Brief Title: Inhaled Polymyxin E to Prevent VAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, doctor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025VAP
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Ventilator-Associated Pneumonia (VAP); Inha'le'd
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NS Group (Placebo Comparator): The patients began to nebulize the drugs within 24 hours after screening. Both groups inhaled twice a day for 3 days. The NS group inhaled with normal saline .
  Interventions: Drug: Inhaled Placebo
- Polymyxin E Group (Experimental): The patients began to inhaled the drugs within 24 hours after screening. Both groups inhaled twice a day for 3 days. The Polymyxin E Group inhaled polymyxin E 75 mg bid .
  Interventions: Drug: inhaled corticosteroids and other asthma drugs

INTERVENTIONS:
Drug: Inhaled Placebo — Inhalation of drugs was started within 24 hours after the screening of patients. Both groups inhaled with vibrating mesh spray twice a day for 3 days. The NS group inhaled with normal saline .
  Arms: NS Group
Drug: inhaled corticosteroids and other asthma drugs — Inhalation of drugs was started within 24 hours after the screening of patients. Both groups used vibrating mesh spray twice a day for 3 days. The Polymyxin E group inhaled polymyxin， 75 mg bid.
  Other Names: Inhaled
  Arms: Polymyxin E Group

SUMMARY:
Ventilator associated pneumonia is the most common manifestation of hospital acquired infections in ICU. The incidence of ventilator-associated pneumonia in patients receiving mechanical ventilation is as high as 20% -71%, which can lead to increased systemic antibiotic use, prolonged mechanical ventilation time and ICU stay, and increased treatment costs. In addition, ventilator-associated pneumonia is also the main cause of hospital infection related deaths in critically ill patients.

However, there is a certain buffer time for patients to develop ventilator-associated pneumonia after receiving endotracheal intubation. Previous studies have found that the peak incidence occurs after 7 days of mechanical ventilation, so there is an opportunity for early treatment to prevent infection. Despite the implementation of numerous preventive measures for ventilator-associated pneumonia over the decades, such as reducing sedation and withdrawal protocols, patient positioning, oral care, prophylactic probiotics, prophylactic antibiotics, and the use of silver plated endotracheal tubes. Among them, the research on the preventive use of antibiotics has a history of over 30 years and is a topic of substantial debate. Prophylactic use of antibiotics includes systemic application and local nebulization inhalation, and inhaled antibiotics may be an effective measure for preventing ventilator-associated pneumonia. Potential extensively drug-resistant Gram negative (XDR-GN) bacteria, such as Escherichia coli, Klebsiella pneumoniae, Pseudomonas aeruginosa, and Acinetobacter baumannii, are common pathogens causing VAP in ICU. The mortality rate of VAP caused by XDR-GN pathogen may be higher than 70%. With the increasing incidence of multidrug-resistant microorganisms, nebulized or inhaled aminoglycoside antibiotics are often used as empirical or definitive treatment for VAP in ICU patients. The previous group of antibiotics, polymyxin, has returned to the view of medical staff. Sodium polymyxin E methanesulfonate has been used as a salvage therapy for XDR-GN bacteria causing pneumonia, demonstrating its activity against XDR-GN causing VAP in critically ill patients. The guidelines of the Infectious Diseases Society of America (IDSA) on hospital acquired pneumonia also indicate that patients with Gram negative pneumonia caused by drug-resistant bacteria are sensitive to polymyxins. In this randomized controlled study, we aim to investigate the effect of prophylactic use of polymyxin E nebulized inhalation on the incidence of VAP.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Patients with brain injury admitted to ICU (including brain injury caused by trauma, cerebral hemorrhage, cerebral infarction, and cardiac arrest)
3. GCS score<12 points
4. Mechanical ventilation time ≥ 48 hours
5. Sign informed consent

Exclusion Criteria:

1. Existing lung diseases that require long-term inhaled medication treatment.
2. Lower respiratory tract infection at admission.
3. New or persistent infiltration on chest imaging within 48 hours after admission.
4. Expected removal of endotracheal tube within the next 24 hours.
5. Mechanical ventilation time before enrollment exceeds 96 hours.
6. Tracheostomy patients.
7. Current or recent use of polymyxin E (within 24 hours).
8. Allergy to polymyxin E.
9. Allergic pregnant or lactating women.
10. Severe neuromuscular lesions.
11. Severe other organ dysfunction. Expected short-term death (48 hours) or palliative treatment.
12. Late stage solid organ or blood system tumors. Expected survival<30 days. 13. Participate in other clinical studies within 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of VAP | From randomization to 7 days
  The incidence of VAP from randomization to day 7.

SECONDARY OUTCOMES:
VAP incidence within 28 days | From randomization to 28 days
  Incidence of VAP from randomization to day 28
Changes of CPIS within day 28 | from randomization to extubation or day 28, whichever occurs first
  Changes of clinical pulmonary infection scores after randomization（CPIS）
Use of systemic antibiotic | From randomization to day 28
  The number of days of systemic antibiotic use and the daily dose of antibiotics administered within 28 days after randomization.
Success of SBT | From randomization to first success of SBT
  The number of days from randomization to the first successful spontaneous breathing test（SBT）
Invasive ventilator-free days at 28 days | From randomization to 28 days
  Days alive without endotracheal intubation and invasive mechanical ventilation
Successful of weaning from ventilator | From randomization to 28 days
  The proportion of patients who Successfully weaned from mechanical ventilator within 28 days.
ICU days at day 28 | From randomization to 28 days
  The number of ICU days within 28 days after randomization
Hospital days at day 28 | From randomization to 28 days
  The number of Hospital days within 28 days after randomization
28-day mortality | From randomization to 28 days
  The proportion of patients who are died within 28 days
Incidence of AKI | From randomization to day 28
  The proportion of patients who were newly diagnosed AKI within 28 days after randomization

IPD SHARING:
Plan to Share IPD: No